CLINICAL TRIAL: NCT05529316
Title: A Multicohort, Open Label, Phase 2 Study of Botensilimab (AGEN1181) for Treatment of Advanced Melanoma Refractory to Prior Checkpoint Inhibitor Therapy
Brief Title: A Study of Botensilimab (AGEN1181) for the Treatment of Advanced Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-800-23; 2022-500652-37 (EudraCT Number)
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Advanced Melanoma
Keywords: Open-label; Monotherapy; Combination Therapy; Anti-PD-1; Anti-PD-L1; Anti-CTLA-4; Immunotherapy
MeSH Terms: interventions — balstilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 Cohort A: Botensilimab (Experimental): Participants refractory to PD-(L)1 therapy will receive botensilimab intravenously (IV).
  Interventions: Drug: Botensilimab
- Part 1 Cohort B: Botensilimab (Experimental): Participants refractory to PD-(L)1 and anti-CTLA-4 therapies will receive botensilimab IV.
  Interventions: Drug: Botensilimab
- Part 2 Cohort A: Botensilimab + Balstilimab (Experimental): Participants refractory to PD-(L)1 will receive botensilimab IV in combination with balstilimab IV.
  Interventions: Drug: Botensilimab; Drug: Balstilimab
- Part 2 Cohort B: Botensilimab + Balstilimab (Experimental): Participants refractory to PD-(L)1 and CTLA-4 will receive botensilimab IV in combination with balstilimab IV.
  Interventions: Drug: Botensilimab; Drug: Balstilimab

INTERVENTIONS:
Drug: Botensilimab — An anti-CTLA-4 monoclonal antibody
  Other Names: AGEN1181
Drug: Balstilimab — An anti-PD-1 monoclonal antibody
  Other Names: AGEN2034
  Arms: Part 2 Cohort A: Botensilimab + Balstilimab; Part 2 Cohort B: Botensilimab + Balstilimab

SUMMARY:
This study is an open-label, 2-part, Phase 2, multicenter study to evaluate the efficacy, safety, tolerability, and pharmacokinetic profiles of botensilimab as monotherapy and in combination with balstilimab in participants with advanced cutaneous melanoma refractory to checkpoint inhibitor therapy.

DETAILED DESCRIPTION:
This Phase 2 study will enroll up to approximately 220 evaluable adult participants with a histologically confirmed diagnosis of either Stage III (unresectable) or Stage IV cutaneous melanoma and who have had prior treatments with anti-programmed death (ligand) 1 [PD-(L)1].

This study will consist of 2 parts. Part 1 consists of 2 cohorts (Cohorts A and B) that will receive botensilimab monotherapy. In Cohort A, participants refractory to PD-(L)1 will receive botensilimab. In Cohort B, participants refractory to PD-(L)1 and cytotoxic T-lymphocyte antigen 4 (CTLA-4) will receive botensilimab. Part 2 consists of Cohorts A and B that will receive botensilimab combination therapy. In Cohort A, participants refractory to PD-(L)1 will receive botensilimab in combination with balstilimab. In Cohort B, participants refractory to PD-(L)1 and CTLA-4 will receive botensilimab in combination with balstilimab.

ELIGIBILITY:
Inclusion Criteria:

To participate in the study, participants must meet all the following inclusion criteria:

Cohort A only:

1. Prior treatment with anti-PD-(L)1 therapy (for example, pembrolizumab or nivolumab) for at least 6 weeks and radiologic progression confirmed by 2 scans at least 4 weeks apart, or if symptomatic due to progressive malignancy, then 1 scan showing progression is sufficient.
2. Progression must be either on treatment with anti-PD-(L)1 regimen or ≤ 12 weeks from last anti-PD-(L)1 dose in metastatic setting or ≤ 24 weeks from completion of therapy in adjuvant/ neoadjuvant setting.
3. For Part 2 only, no intervening anti-cancer therapy between the last course of anti-PD-(L)1 treatment and the first dose of study treatment except for local measures (for example, surgical excision, biopsy, focal radiation therapy), or BRAF ± MEK inhibition when applicable in BRAF mutant participants.

Cohort B only:

1. Prior treatment with first-generation anti-CTLA-4 therapy (for example, ipilimumab or tremelimumab) and prior treatment with anti-PD-(L)1 for at least 6 weeks.
2. Progression on most recent anti-cancer therapy.
3. For Part 2 only, no more than 3 prior lines of therapy in the advanced setting for BRAF mutant and no more than 2 prior lines of therapy in the advanced setting in the BRAF wild type.

Cohorts A and B:

1. Voluntarily agree to participate by giving signed, dated, and written informed consent prior to any study-specific procedures.
2. Histologically confirmed Stage III (unresectable) or Stage IV histologically confirmed cutaneous melanoma as per the American Joint Committee on Cancer 8th edition staging system.
3. Measurable disease on baseline imaging per RECIST 1.1 criteria.
4. BRAF V600 mutation status or consent to BRAF V600 mutation testing per local institutional standards during the screening period.
5. Life expectancy ≥ 3 months.
6. Eastern Cooperative Oncology Group performance status of 0 or 1.
7. Adequate organ function is defined as the following laboratory values within 14 days of Cycle 1 Day 1 (C1D1):

   1. Neutrophils > 1500/microliter (μL) (stable off any growth factor within 4 weeks of first study treatment administration).
   2. Platelets > 100 × 10^3/μL (transfusion to achieve this level is not permitted within 2 weeks of first study treatment administration).
   3. Hemoglobin > 8.0 grams/deciliter (g/dL) (transfusion to achieve this level is not permitted within 2 weeks of first study treatment administration).
   4. Creatinine clearance ≥ 45 milliliters/minute (measured or calculated using modification of diet in renal disease).
   5. Aspartate aminotransferase/alanine aminotransferase < 3.0 × upper limit of normal (ULN).
   6. Total bilirubin < 1.5 × ULN, or < 3.0 × ULN for participants with Gilbert syndrome.
   7. Albumin ≥ 3.0 g/dL.
   8. International normalized ratio or prothrombin time ≤ 1.5 × ULN and activated partial thromboplastin time ≤ 1.5 × ULN (unless participant is receiving anticoagulant therapy).
8. Participant must provide a formalin-fixed paraffin-embedded tumor tissue sample from the most recent biopsy of a tumor lesion, obtained within 90 days from signing informed consent form. If recent tumor tissue is unavailable or inadequate, a fresh biopsy will be required, unless the Sponsor agrees that it is not safe/feasible.
9. Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test at screening (within 72 hours of first dose of study medication) and prior to study drug administration. In part 1, WOCBP must agree to use highly effective contraceptive measures starting with the screening visit through 3 months after the last dose of study treatment. In Part 2, WOCBP must agree to use highly effective contraceptive measures starting with the screening visit through 5 months after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the participant.
10. In Part 1, male participants with a female partner(s) of childbearing potential must agree to use highly effective contraceptive measures throughout the study, starting with the screening visit through 3 months after the last dose of study treatment is received. In Part 2, male participants with a female partner(s) of childbearing potential must agree to use highly effective contraceptive measures throughout the study starting with the screening visit through 5 months after the last dose of study treatment is received. Males with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.

Exclusion Criteria:

To participate in the study, participants must meet none of the following exclusion criteria:

Cohort A:

1. Received prior anti-CTLA-4 therapy.

Cohort B:

1. Received prior Fc-engineered or Fc-enhanced anti-CTLA-4 therapy (for example, BMS-96218, BMS-986288, HBM4003, XTX101, CTLA-4 targeting bispecific or other approaches such as ONC-392).

Cohorts A and B:

1. Ocular, uveal, or mucosal melanoma.
2. Any persistent toxicities (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≥ 2) from prior cancer therapy, excluding endocrinopathies stable on medication, stable neuropathy, and alopecia.
3. Any history of CTCAE Grade ≥ 3 immune-mediated toxicity (excluding endocrinopathies and non-necrotizing/bullous rash) from prior checkpoint inhibitor therapy that required treatment with systemic corticosteroids (> 10 mg/day prednisone or equivalent) or other immunosuppressive medications for more than 4 weeks.
4. Refractory ascites require 2 or more therapeutic paracentesis in the last 4 weeks or ≥ 4 within the last 90 days prior to study entry.
5. Bowel obstruction within the past 3 months or an impending bowel obstruction.
6. Clinically significant (that is, active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥ III), or serious uncontrolled cardiac arrhythmia requiring medication.
7. Active brain metastases or leptomeningeal metastases with the following exceptions:

   1. Treated brain metastases require a) surgical resection, or b) stereotactic radiosurgery. These participants must be off steroids ≥ 10 days prior to randomization for the purpose of managing their brain metastases. Repeat brain imaging following surgical resection or stereotactic radiosurgery is not required if their last brain magnetic resonance imaging is within screening window. Whole-brain radiation is not allowed.
   2. Untreated isolated brain metastases that are too small for treatment by surgical resection or stereotactic radiosurgery (for example, 1-2 millimeters) and/or of uncertain etiology are potentially eligible but need to be discussed with and approved by the study Medical Monitor.
8. Concurrent malignancy (present during screening) requiring treatment or history of prior malignancy active within 2 years prior to the first dose of study treatment (that is, participants with a history of prior malignancy are eligible if treatment was completed at least 2 years before the first dose of study treatment and the participant has no evidence of disease). Participants with history of prior early-stage basal/squamous cell skin cancer, low-risk prostate cancer eligible for active surveillance or noninvasive or in situ cancers who have undergone definitive treatment at any time are also eligible.
9. Incomplete resolution of clinically significant adverse events related to most recent therapy/intervention prior to enrollment.
10. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccine or booster < 7 days before C1D1. For vaccines requiring more than 1 dose, the full series should be completed prior to C1D1, when feasible. A booster shot is not required but if given, must be administered > 7 days from C1D1 or > 7 days from future cycle on study.
11. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
12. Any evidence of current interstitial lung disease (ILD) or pneumonitis or a prior history of ILD or non-infectious pneumonitis requiring high-dose glucocorticoids.
13. History of allogeneic organ transplant, stem cell transplant or bone marrow transplant (autologous stem cell transplant > 5 years prior to study enrollment with no evidence of disease are eligible unless lymphopenia Grade > 1 is present).
14. Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
15. Participants with a condition requiring systemic treatment with either corticosteroids (> 10 milligrams [mg] daily prednisone equivalent) within 14 days or another immunosuppressive medication within 30 days of the first dose of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
16. Active autoimmune disease or history of autoimmune disease that required systemic treatment within 2 years before starting study treatment (that is, with use of disease-modifying agents or immunosuppressive drugs).
17. History or current evidence of any condition, co-morbidity, therapy, any active infections, or laboratory abnormality that might confound the results of the study, interfere with the participants participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating Investigator.
18. A WOCBP who is pregnant or breastfeeding or WOCBP who are not willing to employ effective birth control from screening to 90 days after the last dose of botensilimab (whichever is later).
19. Previous SARS-CoV-2 infection within 10 days for mild or asymptomatic infections or 20 days for severe/critical illness prior to C1D1.
20. Uncontrolled infection with human immunodeficiency virus (HIV). Participants on stable highly active antiretroviral therapy with undetectable viral load and normal cluster of differentiation 4 counts for at least 6 months prior to study entry are eligible. Serological testing for HIV at screening is not required.
21. Known to be positive for hepatitis B virus (HBV) surface antigen, or any other positive test for HBV indicating acute or chronic infection. Participants who are receiving or who have received anti-HBV therapy and have undetectable HBV DNA for at least 6 months prior to study entry are eligible. Serological testing for HBV at screening is not required.
22. Known active hepatitis C virus (HCV) as determined by positive serology and confirmed by polymerase chain reaction (PCR). Participants on or who have received antiretroviral therapy are eligible, provided they are virus-free by PCR for at least 6 months prior to study entry. Serological testing for HCV at screening is not required.
23. Dependence on total parenteral nutrition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | First dose through up to 3 months
  Objective response rate will be determined using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Progression-free Survival | From first dose to first observation of documented disease progression (or death within 12 weeks of last tumor assessment) (up to 3 months)
  Progression-free survival will be determined using RECIST 1.1.
Duration Of Response | From first dose to first observation of documented disease progression (or death within 12 weeks of last tumor assessment) (up to 3 months)
  Duration of response will be determined using RECIST 1.1.
Overall Survival Time | First dose through up to 3 months
  Overall survival will be quantified as a median.
Frequency of Treatment-emergent Adverse Events | First dose through up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Agenus Inc.
Locations (51):
- United States (7):
  - Scottsdale Healthcare Hospitals DBA HonorHealth, Scottsdale, Arizona
  - Virginia K. Crosson Cancer Center at St. Jude Medical Center, Fullerton, California
  - Providence Saint John's Health Center, Santa Monica, California
  - Yale University School of Medicine - Yale Cancer Center, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
- Universitair Ziekenhuis Brussel, Jette, Belgium
- Brazil (7):
  - Oncosite - Centro de Pesquisa Clinica Em Oncologia, Ijuí
  - Centro de Pesquisas Clinicas da Fundação Doutor Amaral Carvalho, Jaú
  - Centro Gaucho Integrado de Oncologia, Hematologia, Ensino e Pesquisa, Porto Alegre
  - INCA II - Instituto Nacional de Cancer Jose Alencar Gomes da Silva, Rio de Janeiro
  - Hospital Sirio Libanes, São Paulo
  - Real e Benemerita Associaçao Portuguesa de Beneficencia - A Beneficencia Portuguesa de Sao Paulo, São Paulo
  - Hospital A.C. Camargo Cancer Center, São Paulo
- France (7):
  - CHU Amiens Picardie - Hopital Sud, Amiens
  - CHU Grenoble-Alpes - Hopital Michallon, La Tronche
  - Centre Leon Berard, Lyon
  - CHU de Nantes, Nantes
  - AP-HP Hopital Saint-Louis, Paris
  - Centre Eugene Marquis, Rennes
  - Gustave Roussy, Villejuif
- Germany (8):
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - University Hospital Schleswig-Holstein, Kiel
  - Universitaetsmedizin der Johannes Gutenberg - Universitaet Mainz, Mainz
  - Klinikum der Universitaet München, München
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaetsklinikum Würzburg, Würzburg
- Italy (3):
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori Dino Amadori - IRST S.r.l., Meldola
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - Azienda Ospedaliero Universitaria Senese, Siena
- Russia (6):
  - Blokhin National Medical Research Oncology Centre, Moscow
  - Branch Office of "Hadassah Medical Ltd", Moscow
  - Moscow City Oncology Hospital #62, Moscow
  - LLC Medical Services, Saint Petersburg
  - Clinical Hospital Russian Railways - Medicine, Saint Petersburg
  - Petrov National Medical Research Center of Oncology, Saint Petersburg
- Spain (7):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Onkologikoa, Donostia / San Sebastian
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Consorcio Hospital General Universitario de Valencia, Valencia
- Switzerland (2):
  - CHUV - Centre hospitalier universitaire vaudois, Lausanne
  - Universitaetsspital Zuerich, Zurich
- United Kingdom (3):
  - Royal Marsden Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Mount Vernon Cancer Centre, Middlesex